CLINICAL TRIAL: NCT03930095
Title: A Randomized Clinical Trial of an Acceptance-based Behavioral Therapy With Mindfulness and Exposure Interventions for Generalized Anxiety Disorder
Brief Title: Efficacy of an Acceptance-based Group Behavioral Therapy for Generalized Anxiety Disorder.
Acronym: ABBT-GAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 51363615.4.0000.0068
Record Dates: First submitted 2019-04-15; First posted 2019-04-29 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2019-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This was a controlled randomized clinical trial involving 10 sessions of ABBT or 10 sessions of NDST (both in groups) completed within 14 weeks.
Who Masked: Participant
Masking Description: After all the participants signed a consent form, each subject was randomized to a single treatment by using the method of randomly permuted blocks (Matts & Lachin, 1988) on http://www.randomization.com. Randomization was stratified in two blocs by use of psychotropic medication in order to have medication use equally distributed between groups. To that end, patients on psychotropic medication were randomized first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance-Based Behavior Therapy (Experimental): 10 sessions of a two-hour group therapy with 12 participants during 14 weeks
  Interventions: Behavioral: Acceptance-based Behavior Therapy
- Non-directive Supportive Therapy (Active Comparator): 10 sessions of a two-hour group therapy with 12 participants during 14 weeks
  Interventions: Behavioral: Non-directive Supportive Therapy

INTERVENTIONS:
Behavioral: Acceptance-based Behavior Therapy — The protocol is widely based on Roemer and Orsillo (2007) acceptance model of GAD, using functional assessment, psychoeducation, mindfulness, commitment to valued behavior, and exposure techniques used in a willingness improvement verbal context.
  Other Names: ABBT; Mindfulness-based Behavior Therapy
  Arms: Acceptance-Based Behavior Therapy
Behavioral: Non-directive Supportive Therapy — NDST consists in a form of therapeutic intervention from which all intervention principles pertaining to specific psychotherapeutic protocols are removed while maintaining the so-called common factors from different psychotherapy approaches. In other words, it is an unstructured therapy without specific psychological techniques other than those belonging to the basic interpersonal skills of the therapist, such as reflection, empathic listening, encouragement, and helping people to explore and express their experiences and emotions.
  Other Names: NDST; Supportive Therapy
  Arms: Non-directive Supportive Therapy

SUMMARY:
Generalized anxiety disorder (GAD) shows the weakest treatment response among anxiety disorders. The present study aimed at examining whether an acceptance-based behavioral treatment, combining mindfulness and exposure strategies, would improve clinical outcome compared to a standard, non-directive, supportive group therapy (NDST) for clients at a Brazilian anxiety disorders program.

DETAILED DESCRIPTION:
Ninety-two individuals diagnosed with GAD were randomized to receive 10 sessions of either an acceptance-based behavior therapy (ABBT) or a Non-directive support Therapy (NDST). Assessments were at pretreatment, mid term, post-treatment, and 3-month follow-up.Data were analyzed using the Mixed effect regression models comparing both groups in primary outcome measures. Secondary outcome measures and putative process variables were assessed and also analyzed. The latter were tested as mediators of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Literate,
* GAD-diagnosed
* 18-65 years old

Exclusion Criteria:

* Bipolar disorder (or any past maniac episodes),
* Psychosis,
* Substance dependence (apart from those abstemious for 3 months or more, considered as initial remission by DSM 5 - APA, 2015),
* High suicide risks according to the MINI - International Neuropsychiatric Interview (MINI; Sheehan et al., 1998).
* Participants under pharmacological treatment for GAD whose medication dosage had not been stable for a minimum of three months prior to the beginning of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2016-08-06 (Actual); Study Completion 2016-08-06 (Actual)

PRIMARY OUTCOMES:
Change in the Depression, Anxiety and Stress Scales | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The 21-item version (DASS-21; Lovibond e Lovibond, 1995), which measures the scores of depression, anxiety and stress separately (7-items each). We followed Roemer & Orsillo (2008) in this study by using the anxiety and stress subscales as general signs of anxiety. Higher scores indicate higher severity of symptoms. Scores are between 0 and 42 for each one of the three subscales. The cut-off scores for conventional severity labels (normal, mild, moderate, severe, extremely severe) are as follows: Anxiety (0-7; 8-9; 10-14; 14-19; 20+) and Stress (0-14; 15-18; 19-25; 26-33; 34+).
Change in the Hamilton Anxiety Scale | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The Hamilton Anxiety Scale (Hamilton, 1959, The assessment of anxiety states by rating) was used to measure anxiety symptoms. The HAM-A is a 14-item interview-administered measure of anxiety widely used in clinical trials, being required as an inclusion criterion in meta-analyses of psychological treatments for anxiety disorders (Bandelow, 2015). Higher scores indicate higher levels of anxious symptoms. The internal consistencies for the HAM-A were .84, .81, .80, and .86 across the four time points. The score ranges from 0 to 54.
Change in the Penn State Worry Questionnaire (Meyer, 1990) | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  it is a 16-item 5-points likert questionnaire with items ranging from 1 (not at all typical of me) to 5 (very typical of me) that measures the trait levels of worry. the scale ranges from 16 to 80. Higher scores indicate higher levels of worry.Its internal consistencies in the current sample were .91, .89, .90, and .92 across the four time points.
Change in the Clinical Global Impressions (CGI; Guy, 1976) | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.The CGI actually comprises two companion one-item measures evaluating the following: (a) severity of psychopathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale (Busner & Targum, 2007). Higher scores indicate higher severity of symptoms or worse evolution.

SECONDARY OUTCOMES:
Change in the Depression sub scale of Depression, Anxiety and Stress Scales | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The 21-item version (DASS-21; Lovibond e Lovibond, 1995), which measures the scores of depression, anxiety and stress separately. We applied the depression factor as a secondary outcome measure. Higher scores indicate higher severity of symptoms. Scores are between 0 and 42. The cut-off scores for conventional severity labels (normal, mild, moderate, severe, extremely severe) for the depression sub scale is (0-9, 10-13, 14-20, 21-27, 28+)
Change in the abridged version of the quality of life inventory - World Health Organization Quality of Life ( WOQOL-BREF - Berlim, Pavanello, Caldieraro, & Fleck, 2005) | Pre-treatment (week 0) one week before the first group session (week 1); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The WHOQOL-BREF is a 26-item questionnaire which includes one item from each of the 24 facets contained in the WHOQOL-100 and two additional items on overall quality of life and general health. The 24 items are organized into 4 domains, namely Physical Health, Psychological, Social Relationships and Environment. In this study we analysed only the fis=rst three domains, because environment characteristics was not supposed to change with psychological interventions. The internal consistencies for WHOQOL were .77, .77, and .81 for the psychological subscale, .78, .76, and .82, for the physical subscale, and .72, .64, and .73 for the social subscale across pretreatment, posttreatment, and 3 month follow up. Higher scores indicate higher quality of Life. Scores of physical, psychological and social domains range from 7 to 35; 6 to 30 and 3 to 15.
Change in the Sheehan Disability Scale (Sheehan, Harnett-Sheehan, & Raj, 1996) | Pre-treatment (week 0) one week before the first group session (week 1); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  It is a discretized analog disability scale (DISS) which uses visual-spatial, numeric and verbal descriptive anchors to assess disability across three domains: work, social life and family life. The internal consistencies for the Sheehan were .71, .80, and .91 across pretreatment, posttreatment, and 3 month follow up. Higher scores indicate higher disability. Scores range from 1 to 10 for each domain.
Change in the Acceptance and Action Questionnaire score | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The Acceptance and Action Questionnaire (AAQ-II-7: Bond, 2011; Flederus, 2012) is a 7-item uni-dimensional measure that assesses experiential avoidance: the unwillingness to remain in contact with aversive private experience and behaviors aimed at altering these experiences or the events that elicit them. Items are scored on a 7-point likert scale ranging from 1 (never true) to 7 (always true). Higher scores indicate higher levels of experiential avoidance and lower levels of psychological flexibility
Change in the Five Facets of Mindfulness Questionnaire score | Pre-treatment (week 0) one week before the first group session (week 1); intermediate assessment (midterm) in the sixth session (week 6); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26)
  The 39-items Five Facets of Mindfulness Questionnaire (FFMQ; Baer et. al., 2006, adapted for Brazil by Barros, 2014), was used for measuring mindfulness in a multidimensional manner for a factorial analysis of different elements of the construct, divided in five domains (i.e. observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience). Items are scored on a 5-point likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Higher scores indicate higher levels of mindfulness.
Change in the Credibility and Expectancy Questionnaire score | This scale was administered at the end of each therapy session throughout the entire treatment.
  The Credibility and Expectancy Questionnaire (CEQ; Borkovec & Nau, 1972; Devilly & Borkovec, 2000) is a 6-item self-report instrument that measures treatment credibility and client expectancy for improvement. The first four items of this scale (set I) are rated based on cognitive appraisal whereas the last two items (set II) are rated based on feelings about the therapy. One item of each set is scored as porcentage (0 to 100) and all of the other items are scored on a 9-point likert scale ranging from 1 (nota t all) to 9 (very). Higher scores indicate higher levels of credibility (first 3 items) and expectancy (last 3 items).
Change in the Mental Health Continuum - Short Form - score | Pre-treatment (week 0) one week before the first group session (week 1); the post-treatment assessment occurred on the day of the tenth session (week 14); and follow-up (week 26
  The MHC-SH (Keyes, 2009 - adapted to Brazilian population by Machado and Bandeira, 2015 ) is a 14-item self-responding instrument that measures positive mental health, witch is understood as symptoms of good affection, self development and social connectivity. Items are scored on a 6-point likert scale ranging from 1 (never) to 6 (every day). The score ranges from 14 to 84. Higher scores indicate higher levels of mental health.
Change in serum C-Reactive Protein (CRP) | Before the first session (week 1) and after the last session (week 14)
  Blood samples were collected before and after psychological interventions. High sensitivity CRP, expressed in mg/L, was measured using immunoturbidimetric method. High scores indicate cardiovascular risk and/or presence of infectious or inflammatory processes.
Change in serum inflammatory markers | Before the first session (week 1) and after the last session (week 14)
  Blood samples were collected before and after psychological interventions. Serum levels of IL-1beta, IL-4, IL-6, IL-8, IL-10, TNFalpha and Vascular Endothelial Growth Factor (VEGF), all expressed in pg/mL, were quantified simultaneously using Luminex xMAP technology with a commercial multiplex immunoassay kit according to the manufacturer's instruction.
Change in Brain Derived Neurotrophic Factor (BDNF) plasma levels | Before the first session (week 1) and after the last session (week 14)
  Blood samples were collected before and after psychological intervention. Plasma levels of BDNF were measured using an enzyme-linked immunosorbent assay (ELISA).
Change in serotonin plasma levels | Before the first session (week 1) and after the last session (week 14)
  Blood samples were collected before and after psychological intervention. Plasma levels of serotonin were measured using an enzyme-linked immunosorbent assay (ELISA).
Change in the Temperament and Character Inventory - Revised (TCI-R) scores | Pre-treatment (week 0) and after the last session (week 14)
  The TCI-R is a self-reported questionnaire, with 240 questions that require answers in a 5-point-Likert scale. Each question is related to one of the seven factors described by the authors of the scale: novelty seeking, harm avoidance, reward dependence, persistence, self-directedness, cooperativeness and self-transcendence.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Lotufo Neto, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Department and Institute of Psychiatry - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No